CLINICAL TRIAL: NCT04498286
Title: COVID-19 and SARS-CoV-2 Antibodies in Multiple Sclerosis Patients: a Large Study in the Amsterdam MS Cohort
Brief Title: COVID-19 and SARS-CoV-2 Antibodies in Multiple Sclerosis Patients
Acronym: COMS-19
Status: Completed | Type: Observational
Sponsor: Zoé van Kempen (Other)
Responsible Party: Sponsor-Investigator, Zoé van Kempen, PhD, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Other Study IDs: NL74243.029.20
Record Dates: First submitted 2020-08-03; First posted 2020-08-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amsterdam MS Cohort
  Interventions: Diagnostic Test: Testing of SARS-CoV-2 antibodies

INTERVENTIONS:
Diagnostic Test: Testing of SARS-CoV-2 antibodies — Sars-CoV-2 RBD total antibody test developed by Sanquin

SUMMARY:
Rationale: Patients with MS are possibly more vulnerable to infection with SARS-CoV-2. Furthermore the use of immunomodulatory treatment could have an effect on the course of COVID-19 disease. This has resulted in an alteration of current immunomodulatory treatment strategies and delaying the start of certain medications, which could induce MS disease activity. However, certain immunomodulatory treatments are also hypothesized to have a positive effect on COVID-19 disease. Besides lack of information regarding the effects of MS treatments on COVID-19, there is significant uncertainty in how we should advise MS patients in terms of self-isolation, resulting in many patients staying at home reluctant to perform their work or other daily activities. Nationally and locally, we are collecting information regarding COVID-19 in MS patients but numbers are low and only those who are severely affected are tested. Furthermore, there is no information regarding SARS-CoV-2 immunity in MS patients, which could be affected by certain MS treatments. Consequently, there is an urgent need for reliable information about infection rates/immunity and course of COVID-19 in relation to MS characteristics and treatments.

Objectives: The objectives of this study are 1. to study the course of COVID-19 in MS patients in relation to immunomodulatory treatment and other patient and MS characteristics and 2. to study the proportion of MS patients with SARS-CoV-2 antibodies and 3. to establish the antibody profile in positive tested patients and 4. to study the longitudinal course of these antibody profiles in positive tested patients.

Study design: This is a mono-center cohort study in patients of the MS Center Amsterdam.

Study population: All patients with a diagnosis of MS currently under follow-up in the Amsterdam MS Center.

Intervention (if applicable): Single venous puncture for drawing blood and questionnaire. For a minority of patients (max 25%) who test positive for antibodies we will draw blood a again with questionnaires after six and twelve months.

Main study parameters/endpoints: Course of COVID-19 in MS patients in relation to MS immunomodulatory treatment.

ELIGIBILITY:
Inclusion Criteria:

* a current diagnosis of multiple sclerosis and age ≥18 years.

Exclusion Criteria:

* lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of MS currently under follow-up in the MS Center Amsterdam.
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
The correlation of COVID-19 disease course with MS immunomodulatory treatment | at baseline questionnaires and lab results
  Correlationg of disease course of COVID-19 in patients with positive SARS-CoV-2 antibodies defined by questionnaires (asymptomatic, mild symptoms, severe symptoms, hospitalization) with MS immunomodulatory treatment (asked by questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Zoé L van Kempen, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU medical center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boekel L, Steenhuis M, Hooijberg F, Besten YR, van Kempen ZLE, Kummer LY, van Dam KPJ, Stalman EW, Vogelzang EH, Cristianawati O, Keijzer S, Vidarsson G, Voskuyl AE, Wieske L, Eftimov F, van Vollenhoven R, Kuijpers TW, van Ham SM, Tas SW, Killestein J, Boers M, Nurmohamed MT, Rispens T, Wolbink G. Antibody development after COVID-19 vaccination in patients with autoimmune diseases in the Netherlands: a substudy of data from two prospective cohort studies. Lancet Rheumatol. 2021 Nov;3(11):e778-e788. doi: 10.1016/S2665-9913(21)00222-8. Epub 2021 Aug 6. PMID 34396154